CLINICAL TRIAL: NCT04267757
Title: Transperineal Repair of Primary Obstetric Rectovaginal Fistulas With Fecal Incontinence Using Fistulectomy, Sphincteroplasty and With or Without Bulbocavernosus Muscle Flap:Surgical Pitfalls and Prevention of Recurrence
Brief Title: Transperineal Repair of Primary Obstetric Rectovaginal Fistulas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Tamer Alsaied Alnaimy, assistant professour, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: zagazig 2
Record Dates: First submitted 2020-02-09; First posted 2020-02-13 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Recto Vaginal Fistula
MeSH Terms: conditions — Rectovaginal Fistula

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Experimental): RVF with Martius flap
  Interventions: Procedure: rectovaginal fistula repair with Martius flap
- group 2 (Experimental): RVF without Martius flap
  Interventions: Procedure: rectovaginal fistula repair with Martius flap

INTERVENTIONS:
Procedure: rectovaginal fistula repair with Martius flap — rectovaginal fistula repair with Martius flap

SUMMARY:
Introduction: A rectovaginal fistula (RVF) is an epithelium-lined abnormal tract between the rectum and the vagina and is often a challenging problem for both the patients and to the surgeons. In literature, there is still debate regarding the best treatment options for rectovaginal fistulas.

Aim: To assess the results of the treatment of rectovaginal ﬁstulas with incontinence and impaired anal tonus using fistulectomy, sphincteroplasty with or without bulbocavernosus muscle (Martius) flap.

Materials and Methods: A total of 22 consecutive patients with simple RVFs were included and assigned to transperineal repair. The patients were divided into two groups , group1: with Martius flap; group2: without Martius flap .Postoperatively, patients were followed up for one year at the outpatient clinic or through telephone interviews with speciﬁc questionnaires to collect information on the status of fecal control, ﬂatus, or fecal leakage from the vagina.

DETAILED DESCRIPTION:
Introduction:

Rectovaginal ﬁstulas represent an often devastating condition in patients and a challenge for surgeons because of their irritating and embarrassing symptoms and high failure rate after repair.Patients with rectovaginal ﬁstulas typically present with complaints of passage of ﬂatus or feces from the vagina with painful skin excoriation.

(1) The most common etiological cause of rectovaginal ﬁstulas is obstetrical trauma. When obstructed labor is unrelieved, the presenting fetal part is impacted against the soft tissues of the pelvis leading to ischemic vascular injury and subsequent tissue necrosis and ﬁstula formation. Other predisposing factors include forceps delivery, midline episiotomy, and third or fourth-degree perineal lacerations.( 2).

Evaluation of a patient with rectovaginal ﬁstula includes a detailed history, examination of the rectum, vagina, and perineal body. The perineal body is often thin or nearly nonexistent in patients with sphincter injuries secondary to obstetrical trauma. Endoanal ultrasonography and pelvic Magnetic Resonance Imaging (MRI) to conﬁrm sphincter injury and may provide valuable information before a planned repair. MR is the modality of choice for disease staging (sensitivity 91%) (3).

( Sagittal T2 MR imaging shows communication between the rectum tumor and the vagina) The experience of the surgeon and the previous attempts at repair are also important factors of the success rate of the operations [4)

There are various operative procedures, such as the advancement ﬂap, sphincteroplasty and ﬁstulectomy, coloanal anastomosis,and gracilis muscle repair to manage rectovaginal ﬁstulas [5].

The choice of the operative technique greatly depends on the status of the ﬁstula and the etiological rationale behind this medical complication [6.].

In this study, we have compared the outcomes of the ﬁstulectomy and sphincteroplasty procedures with or without concomitant bulbocavernosus flap. All patients were incontinent and felt to have impaired anal tonus.

Patients and method:

Study design:

This prospective study involved 22 patients diagnosed with simple rectovaginal fistula from January 2018 to January 2019 at the General surgical department, faculty of medicine Zagazig University, Egypt. This study was approved by the institutional ethics board of our hospital. All patients who participated in the study provided informed consent.

rectovaginal examination, endoanal ultrasonography, and pelvic MRI ﬁndings were collected to assess the extension of the fistula. Colonoscopy was performed in selected patients with severe bowel symptoms such as bloody diarrhea to exclude inflammatory bowel disease. Decisions regarding operations were made cautiously and involved the whole medical team. All cases underwent fistulectomy, sphincteroplasty and with or without bulbocavernosus flap technique.All patients were evaluated for incontinence using Wexner Incontinence Score (WIS) [7) Method of randomization: simple randomization with a balance.

Patient selection:

Inclusion criteria:

1. Rectovaginal fistula caused by obstetric problems
2. Female >20 years

Exclusion criteria:

1. other causes of rectovaginal fistula as Crohn's disease or malignant fistula
2. complex and recurrent fistula

Three patients did not undergo surgery. One because of patient's choice, one because of minimal symptoms and one because fistula healed after medical therapy.

Methods:

Patients were given a mechanical bowel preparation the day before surgery and an enema on the morning of the operation. The patient was placed in the lithotomy position under spinal anesthesia. Antibiotics in the form of third generation cephalosporin and 500 mg of Metronidazole were given.

Sub mucosal lidocain 5% in adrenalized saline at a ratio of 1: 100 000 was injected around the fistula. Surgical excision of the fistula using scalpel was performed. Biopsies of rectal mucosa and the fistula margin were also obtained for pathological evaluation to exclude an underlying Crohn's disease or malignancy. A transverse perineal incision was done. Dissection of the internal sphincter fibers away from the external sphincter fibers was performed, allowing a tension free rectal closure at the fistulous site (Dissection of internal sphincter ﬁ bers from external sphincter ﬁ ber s.). Closure of the fistulous opening at the rectal side was done using Vicryl 3/0 sutures. This was followed by suturing of the rectovaginal septum to the internal sphincteric fibers using Vicryl 3/0 sutures (Suturing of internal sphincter ﬁ bers to the rectovaginal septu m.). The bulbocavernosus muscle flap was harvested from the left side in all patients at its anterior part, preserving the posteroexternal vascular pedicle (Posterior muscle repair), through the same incision, and sutured across the rectum to its counterpart on the other side (Vaginal advancement ﬂ a p.& Fig. 1 a The fistulae are indicated by the two forceps passing through them; b The finger demonstrates the large recto-vaginal orifice) using 2/0 Vicryl sutures. The vaginal flap was advanced at the fistula site and sutured to the perineal skin using Vicryl 3/0 sutures (Preparation of the bulbocavernosus ﬂ a p.& Fig. 3 a, b After a right labial incision, the bulbocavernous muscle and the surrounding fibroadipose tissue were carefully mobilized, avoiding possible damage of the postero-external vascular pedicle& Fig. 4 A subcutaneous tunnel connecting the two incisions was created after transecting superior to the bulbocavernous muscle& Fig. 5 The final set-up with the interrupted absorbable sutures over the vaginal closure after sectioning of the longitudinal vaginal septum. The bulbocavernous muscle is clearly visible after the lay open of the perineovaginal tract).

No suction drain was used. No covering stoma was done. Postoperatively, Soft, stool was provided in the postoperative period at least for two weeks with the help of clear liquid diet, plenty ﬂuid intake, and the use of stool softeners. Oral broad-spectrum antibiotic therapy was given for 3-5 days postoperatively. Sexual activity or any physical activities more strenuous than a slow walk were avoided by the patients for three weeks after the surgery. Follow up period up to one year.

ELIGIBILITY:
Inclusion Criteria:

* 1- Rectovaginal fistula caused by obstetric problems 2- Female >20 years

Exclusion Criteria:

1. other causes of rectovaginal fistula as Crohn's disease or malignant fistula
2. complex and recurrent fistula -

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
rectovaginal fistula repair with or without Martius flap | 1 year
  detect recurrence in rectovaginal fistula repair with or without Martius flap

CONTACTS AND LOCATIONS:
Overall Officials: tamer A. alnaimy, MD, Principal Investigator — Zagazig University
Locations (1):
- Tamer Alsaied Alnaimy, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No